CLINICAL TRIAL: NCT05386953
Title: Intraoperative Normal Saline Administration and Acute Kidney Injury in Patients Undergoing Liver Transplantation: a Retrospective Cohort Study
Brief Title: Intraoperative Normal Saline Administration and Acute Kidney Injury in Patients Undergoing Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Professor, Seoul National University Hospital
Other Study IDs: H-2108-173-1248
Record Dates: First submitted 2022-05-15; First posted 2022-05-24 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: End Stage Liver DIsease; Liver Transplant; Complications; Liver Cirrhosis
MeSH Terms: conditions — End Stage Liver Disease; Liver Cirrhosis | interventions — Saline Solution; Ringer's Lactate; stable plasma protein solution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Balanced group: Patients who received balanced crystalloids of lactated Ringer's solution or plasma solution during liver transplantation surgery
  Interventions: Drug: Balanced crystalloid solution
- Saline group: Patients who received only normal saline during liver transplantation surgery
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Normal saline — Patients received normal saline as a maintenance crystalloid during liver transplantation surgery.
  Groups: Saline group
Drug: Balanced crystalloid solution — Patients received balanced crystalloids such as lactated Ringer's solution or Plasma solution as a maintenance crystalloid during liver transplantation surgery.
  Other Names: Lactated Ringer's solution; Plasma solution
  Groups: Balanced group

SUMMARY:
The investigators attempted to investigate the association of the type of crystalloid administered during liver transplantation with postoperative clinical outcomes. The investigators hypothesized that the greater amount of normal saline or half-saline administered during liver transplantation might be associated with the increased risk of acute kidney injury compared to the balanced crystalloids.

DETAILED DESCRIPTION:
Liver transplantation requires a long operation time and is often associated with a significant amount of surgical bleeding. It is common for the anesthesiologist to infuse large amounts of fluid or blood products due to bleeding, hemodynamic instability, or ascites drainage. Therefore, in the anesthesia for liver transplantation, optimal management of fluid administration is necessary and the choice of the type of crystalloid may affect the prognosis or the incidence of postoperative complications of patients.

The investigators attempted to investigate the association of the type of crystalloid administered during liver transplantation with postoperative clinical outcomes. The investigators hypothesized that the greater amount of normal saline or half-saline administered during liver transplantation might be associated with the increased risk of acute kidney injury compared to the balanced crystalloids.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who underwent living or deceased donor liver transplantation at our tertiary care university hospital between 2004 and 2018

Exclusion Criteria:

* patients with baseline renal dysfunction of hepatorenal syndrome or chronic kidney disease
* missing preoperative serum creatinine value
* missing other baseline or outcome variables
* patients who received retransplantation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients received liver transplantation surgery in a single tertiary care university hospital
Sampling Method: Non-Probability Sample
Enrollment: 1440 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | the first 7 postoperative days
  The investigators defined acute kidney injury by the KDIGO (Kidney Disease Improving Global Outcomes) criteria, which was determined according to the greatest change in serum creatinine level during the postoperative seven days (Stage 1: more than 1.5-fold; stage 2: more than 2-fold; stage 3: more than 3-fold increase of baseline or increase in SCr to ≥ 4.0 mg/dL or the initiation of renal replacement therapy). The most recent SCr level measured before surgery was collected as a baseline value.

SECONDARY OUTCOMES:
Incidence of postoperative hemodialysis | the first month after admission
  the incidence of new-onset postoperative hemodialysis during hospitalization
Early allograft dysfunction | the first 7 postoperative days
  One or more of the following are present within the first 7 postoperative days: total bilirubin ≥ 10 mg/dL, PT (prothrombin time):INR (international normalized ratio)≥ 1.6, or AST (aspartate aminotransferase)/ALT (alanine aminotransferase) > 2000 IU/L
In-hospital mortality | the first month after admission
  all-cause mortality during hospitalization
One-year mortality | one year after transplantation
  all-cause mortality during one year after transplantation
Length of intensive care unit stay | the first month after admission
  Length of intensive care unit stay after transplantation
Length of hospital stay | the first month after admission
  Length of hospital stay after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, MD, PhD, Study Chair — Department of Anaesthesiology and Pain Medicine, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No